CLINICAL TRIAL: NCT03715244
Title: Rate of Postoperative Delirium and Postoperative Cognitive Dysfunction After Spinal Anesthesia With Short-acting Local Anesthetics Compared to General Anesthesia After a Shared Decision Making Process
Brief Title: Rate of Postoperative Delirium and Postoperative Cognitive Dysfunction After Spinal Anesthesia
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia Spies, Head of the Department of Anesthesiology and Operative Intensive Care Medicine (CCM/CVK), Charité - University Medicine Berlin, Charite University, Berlin, Germany
Other Study IDs: PODSPA
Record Dates: First submitted 2018-10-09; First posted 2018-10-23 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Delirium
MeSH Terms: conditions — Delirium | interventions — Anesthesia, Spinal; Anesthesia, General

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Apolipoprotein-E-4, ncounter Neuroinflammation and micro RNA Panel from Multiplex-Genexpressionsanalyses
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Study group 1: n=220 patients for routine data of spinal anesthesia with short-acting local anesthetics
  Interventions: Procedure: Spinal anesthesia with short-acting local anesthetics
- Study group 2: n= 220 patients for routine data of general anesthesia (current standard)
  Interventions: Procedure: General anesthesia (current standard)
- No intervention: Control group postoperative cognitive deficit: n= 90 control subjects aged 18 years or older (without surgery) with a similar health status and age as the study group patients (similar distribution in the American Society of Anaesthesiologists physical status classification and relevant co-morbidities, e.g. diabetes, coronary artery disease, hypertension and hyperlipidemia). The patients are analyzed to correct for learning effects of the cognitive assessment testings in the study groups.

INTERVENTIONS:
Procedure: Spinal anesthesia with short-acting local anesthetics — Spinal anesthesia in patients with duration of surgery < 90 minutes
  Groups: Study group 1
Procedure: General anesthesia (current standard) — General anesthesia in patients with duration of surgery < 90 minutes
  Groups: Study group 2

SUMMARY:
The aim of this investigation is to compare the standard of general anesthesia used in these patients with these short-acting local anesthetics (Chloroprocain (Ampres®) and Prilocain (Takipril®)) for spinal anesthesia as well as to report the patient centered outcome of postoperative delirium and neurocognitive disorder. In accordance to current evidence regarding the occurrence of postoperative delirium and postoperative cognitive deficit, patients are to be screened daily for delirium up to the fifth postoperative day if in hospital, or till the first postoperative day after ambulatory surgery and for neurocognitive disorder 1 year following the surgery. To detect delirium the Nu-DESC (Nursing Delirium Screening Scale) will be used as a validated scoring systems to ensure the highest sensitivity in delirium identification. CANTAB battery will be used for assessment of neurocognitive disorder. This is a neuropsychological testing (computer-based (I-Pad) [Cambridge Neuropsychological Test Automated Battery - CANTAB connect and parameters from the item list], as well as the subjective / by proxy Assessment of Cognitive Limitations. It is essential to perform the appropriate cognitive performance tests not only on operative patients but also on a non-surgical cohort, using currently established models of calculation in postoperative cognitive deficits and a control group generated from non-surgical patients.

DETAILED DESCRIPTION:
A conventional spinal anesthesia with long-acting drugs (such as bupivacaine) can lead to delays in postoperative recovery, mobilization, delays in discharge from recovery room and in ambulatory surgery. Short-acting local anesthetics (Chloroprocain (Ampres®) and Prilocain (Takipril®)) might be beneficial in short duration surgery under spinal anesthesia and could improve patients' acceptance for neuroaxial anesthesia as it might improve early recovery and early mobilization. Time to first oral nutritional intake/postoperative nausea and vomiting (PONV), time to discharge from post-anesthesia recovery unit and time to discharge home after ambulatory operation might be reduced and might reduce incidence of postoperative delirium and neurocognitive disorder after peripheral surgery.

It is planned to retrospectively examine a group of surgical patients for the purpose of a comparative descriptive collective. This comparison collective is required for various questions, in particular influencing factors with regard to the postoperative outcomes delirium, neurocognitive disorder and mortality. Only the routine data is used and no additional surveys are performed on these patients. Inclusion criteria such as the study cohort and additionally the inclusion criterion: Spinal anesthesia with another local anesthetic

ELIGIBILITY:
Study group 1 and 2

Inclusion Criteria:

* Surgical patients at Campus Virchow - Klinikum and Campus Charité Mitte (Charité - Universitätsmedizin Berlin)
* Short, elective procedure (<90 minutes), feasible in spinal anesthesia
* American Society of Anesthesiologists (ASA-Score I to III)
* Age ≥ 18 years
* Informed consent process

Exclusion Criteria:

* Non-consenting patients
* Lack of consent to participate in the study or to store, process and disseminate pseudonymised study data
* Allergy or contraindications to local anesthetics
* Contraindications to spinal anesthesia
* Coagulopathy or therapy with anticoagulants
* Higher grade aortic stenosis
* Anomaly of the spinal cord
* Pre-existing neurological deficit
* Pre-existing neurological disease that severely limits the performance of neurocognitive testing
* Hearing and / or visual disturbances (such as color blindness) or relevant language barrier severely limiting the performance of neurocognitive testing
* Spinal anesthesia with another local anesthetic
* Sole peripheral local anesthesia
* Participation in another prospective intervention study
* Emergency operation
* Pregnancy and breast feeding period

POCD Control group:

Inclusion criteria:

* Male and female patients ages 18-100 years, also controls from the POCD registry (EA1/104/16)
* Healthy volunteers (ASA I) / ASA II + III patients who are not scheduled for surgery next year
* Ability to consent to oral and written information
* Patient education and written consent

Exclusion criteria:

* Operation in the last six months before inclusion in this study
* Lack of consent for the pseudonymised disease data to be stored and shared in this clinical trial
* Lack of readiness to participate in the follow-up examinations and contact to make an appointment
* Patients with a neuropsychiatric condition that limits the performance of neurocognitive testing
* Patients with hearing and / or vision disorders or relevant language barriers that limit the performance of neuro-cognitive testing
* Simultaneous participation in a prospective clinical intervention study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Surgical patients at Campus Virchow - Klinikum and Campus Charité Mitte (Charité - Universitätsmedizin Berlin) with short, elective procedure (<90 minutes), feasible in spinal anesthesia
Sampling Method: Probability Sample
Enrollment: 237 (Actual)
Dates: Start 2019-03-12 (Actual); Primary Completion 2021-11-09 (Actual); Study Completion 2022-07-14 (Actual)

PRIMARY OUTCOMES:
Rate of postoperative delirium | Up to five postoperative days
  Postoperative delirum rate, defined according to Diagnostic and Statistical Manual of Mental Disorders (DSM-V) and/or as ≥ 2 cumulative points in the nursing Delirium Screening Scale (Nu-DESC) and/or a positive Confusion Assessment Method (CAM) Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) score and/or patient chart review that shows descriptions of delirium. The basis is the elevation of the sedation depth with the Richmond Agitation Sedation Scale (RASS).

SECONDARY OUTCOMES:
Perioperative cognitive disturbances | Up to 1 year
  Cognitive disorders are evaluated according to DSM-V (formal cognitive testing, subjective memory sensing and instrumental activities of daily living, ).
MONTREAL COGNITIVE ASSESSMENT (MOCA) | Up to 1 year
  Test performance of the MONTREAL COGNITIVE ASSESSMENT (MOCA) for screening of dementia
Formal cognitive testing | Up to 1 year
  Perioperative changes of damain specific test performance in formal cognitive testing
Postoperative cognitive dysfunction (POCD) | Up to 1 year
  Postoperative cognitive dysfunction (POCD) is measured by computerized Cambridge Neuropsychological Test Automated Battery - CANTAB connect and paper pencil testing and subjective memory sensing.
Duration of delirium | Participants will be followed for the duration of hospital stay, an expected average of 7 days ]
  Diagnostic and Statistical Manual of Mental Disorders (DSM-V) Nursing Delirium Screening Scale (Nu-DESC) Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) Confusion Assessment Method (CAM) Chart Review
Severity of delirium | Participants will be followed for the duration of hospital stay, an expected average of 7 days ]
  Diagnostic and Statistical Manual of Mental Disorders (DSM-V) Nursing Delirium Screening Scale (Nu-DESC), Confusion Assessment Method (CAM) and or Confusion Assessment Method for the Intensive Care Unit (CAM-ICU), Chart Review
Time to mobilization | Up to five postoperative days
Time to first oral nutritional intake | Up to five postoperative days
Time until leaving the recovery room | Up to leaving the recovery room
  Fulfillment of discharge criteria from the recovery room
Time until leaving hospital | Up to five postoperative days
  Fulfillment of discharge criteria from hospital after study procedure
Organ complications according to Clavien | Up to five postoperative days
Autonomy Preference Index (API) | Up to five postoperative days
Questionnaire for shared decision making (PEF-FB-9) | Up to five postoperative days
  Results from PEF-FB-9 are evaluated
Total treatment outcome in terms of quality of life of patients | Up to 1 year
  EQ-5D
Total treatment outcome in terms of functional autonomy of patients | Up to 1 year
  Activities of Daily Living (ADLs) or Instrumental Activities of Daily Living (IADLs)
Intraoperative Neuromonitoring | Up to the end of surgical procedure
Cerobrospinal fluid parameter | Until the end of surgery
  Beta-Amyloid 1-40, beta-Amyloid 1-42, beta-Amyloid Ratio (42/40*10), phospho-TAU, Protein 14-3-3, PRPSc, TAU (Gesamt-Tau) from cerobrospinal fluid for measuring dementia
Apolipoprotein E | Until the end of surgery
  Blood marker Apolipoprotein E for measuring dementia
Multiplex Gene Expression Analysis (Whole Blood) | Until first postoperative day
Antibodies | Until first postoperative day
  Antibody from serum (anti-beta2-adrenergic receptor, anti-muscarinic acetylcholine receptor (M3 / M4), anti-serotonin receptor, anti-dopamine receptor)
Pro and anti-inflammatory markers | Until first postoperative day
  IL-8 from whole blood and IL-6, IL-8 and TGF
Immune cells | Until first postoperative day
  Immune cells from citrate blood
Autophagy of platelets | Until first postoperative day
  Autophagy of platelets from citrate blood
Intracellular pH | Until first postoperative day
  Intracellular pH from citrate blood
Cholinesterases | Until the third postoperative day
Anxiety 1 | Up to 1 year
  Anxiety 1 is measured by Generalized Anxiety Disorder 7 (GAD-7) and Patient Health Questionnaire 9 (PHQ-9)
Anxiety 2 | Up to 1 year
  Anxiety 2 is measured by Amsterdam Preoperative Anxiety and Information Scale (APAIS) and Faces Anxiety Scale (FAS)
Subsequent surgery | Up to 1 year
  Results from subsequent surgery are evaluated
Obstructive Sleep Apnea (OSAS) | Up to 1 year
  Obstructive Sleep Apnea (OSAS) is measured by the STOP-Bang Questionnaire.
Fatigue | Up to 1 year
  Fatigue is monitored by Acute Fatigue Score
Sleep behavior | Up to 1 year
  Sleep behaviour is measured by Insomnia Severity Index (ISI) at baseline, 3 months, 1 year
Sleep behavior | Participants will be followed for the duration of hospital stay, an expected average of 7 days ]
  Sleep behaviour is measured by intraclinical course (immediate perioperative: Richards Campbell Sleep Questionnaire)
Frailty | Participants will be measured at the beginning of the investigation.
  Frailty is measured with a modified frailty score according to Fried´s frailty phenotype assessment
Stress | Up to 1 year
  Stress is monitored by Perceived Stress Questionnaire 20 (PSQ20) and Disstressthermometer without areas
Dose of concomitant medication | Up to 5 postoperative days
  The types of medications used in the management of pain, agitation, and delirium on that day are documented.
Duration of concomitant medication | Up to 5 postoperative days
  The types of medications used in the management of pain, agitation, and delirium on that day are documented.
Time of mechanical ventilation | Participants will be followed for the duration of intensive care unit stay, an expected average of 1 day]
Intensive care unit stay | Participants will be followed for the duration of intensive care unit stay, an expected average of 1 day]
Number of stationary recoveries | Up to 1 year
Visits to doctors and outpatient treatments | Up to 1 year
Number of additional operations | Up to 1 year
Mortality | Up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD, Prof., Study Director — Charite University, Berlin, Germany
Locations (1):
- Department of Anesthesiology and Operative Intensive Care Medicine (CCM/CVK), Charité - Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aldecoa C, Bettelli G, Bilotta F, Sanders RD, Audisio R, Borozdina A, Cherubini A, Jones C, Kehlet H, MacLullich A, Radtke F, Riese F, Slooter AJ, Veyckemans F, Kramer S, Neuner B, Weiss B, Spies CD. European Society of Anaesthesiology evidence-based and consensus-based guideline on postoperative delirium. Eur J Anaesthesiol. 2017 Apr;34(4):192-214. doi: 10.1097/EJA.0000000000000594. PMID 28187050
- [Derived] Kipping V, Kerlin TB, Borchers F, Kulken MF, Schmid M, Ahrend CS, Wiebach J, Piper SK, Wernecke KD, Muller A, Spies CD. Postoperative delirium after short-acting spinal anesthesia and general anesthesia after shared decision-making. J Int Med Res. 2025 Sep;53(9):3000605251363408. doi: 10.1177/03000605251363408. Epub 2025 Sep 13. PMID 40945957